CLINICAL TRIAL: NCT06829667
Title: An Open Label, Single Cohort, Multi-center, Retrospective Study of Suture Tape for Soft Tissue Reconstruction in Patients Suffering From Lateral Ankle Instability
Brief Title: Retrospective Study of Suture Tape for Soft Tissue Reconstruction in Patients Suffering From Lateral Ankle Instability
Status: Enrolling by invitation | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: ART-004
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Lateral Ankle Instability
Keywords: ATFL reconstructive procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Arthrex InternalBrace — Arthrex InternalBrace is composed of a polyethylene/polyester suture tape and knotless bone anchors to provide ligament repair bridging and reinforce ligament strength. There have been conflicting results surrounding the clinical efficacy of its use in lateral ligament reconstruction.

SUMMARY:
This study is intended to be a retrospective chart review of patients with chronic ankle instability who have undergone a lateral ligament reconstructive procedure for ATFL repair (isolated or non-isolated) with suture tape augmentation. Patients that have been treated at any of the participating institutions that have undergone an ATFL reconstruction with Arthrex InternalBrace augmentation who have postoperative hospital or ASC records of safety and effectiveness as measured by adverse events, potential complications, and potential functional outcomes past the 10-week time point will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients between and including the age of 14-75 at the time of surgery
* Patients who were diagnosed with lateral ankle instability by physician clinical assessment
* Patients who underwent an ATFL repair with Arthrex InternalBrace augmentation device (does not require an isolated repair)

Exclusion Criteria:

* Significant secondary procedures done at the time of repair, including significant osteochondral lesions and/or significant microfracture of the talus or tibia that warrant modifying the typical lateral ligament repair post-op rehab protocol. (Minor microfractures and OCD lesions that do not warrant bone debridements, synovectomies, and bone spur removals are allowed)
* Any concomitant orthopedic procedure that will extend the post-op rehabilitation (e.g., casting/immobilization) beyond the routinely prescribed rehab protocol following an ATFL reconstructive procedure.
* Patients undergoing a Calcaneal osteotomy
* Patients with less than 6 weeks follow-up
* Patients with incomplete medical records
* Patients with Worker's Compensation Cases
* Any patient with a history of infection of the ankle predating the ankle repair
* Any orthopedic issue outside of the ankle that the Investigator feels may impede functional endpoint outcome measures.
* Patients who have a medical history that would likely make the patient an unreliable research participant

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 75 subjects underwent an ATFL repair with Arthrex InternalBrace
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate Effectiveness | 12 weeks to last recorded follow-up
  The overall objective of this study is to evaluate the effectiveness and safety of suture tape when used as an augmentation device during surgical reconstruction of ATFL in patients suffering lateral ankle instability.
  The assessment of effectiveness will be measured by the rate of complications as defined by those patients that necessitated a return to the OR, including implant failure, symptomatic implant requiring removal, peri-implant fracture, deep wound infection and foreign body reaction.
Evaluate Safety | 2 weeks to last recorded follow-up
  The overall objective of this study is to evaluate the effectiveness and safety of suture tape when used as an augmentation device during surgical reconstruction of ATFL in patients suffering lateral ankle instability.
  Safety of study subjects will be established by recording treatment, incidence and frequency of adverse events. Also, adverse events will be classified as procedure related and/or product related.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma & Extremities
Locations (4):
- United States (4):
  - MORE Foundation, Phoenix, Arizona
  - KUMC, Kansas City, Kansas
  - Seaview Orthopaedics, Ocean City, New Jersey
  - ERLANGER, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No
Unknown at this time